CLINICAL TRIAL: NCT05003570
Title: Efficacy and Safety of Remifentanil for Mechanically Ventilated Patients in Intensive Care: Multicenter, Random, Double-blind, Parallel, Positive Control Clinical Trials
Brief Title: Efficacy and Safety of Remifentanil for Mechanically Ventilated Patients in ICU
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Ling Liu, professor, Southeast University, China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZDRF
Record Dates: First submitted 2021-06-30; First posted 2021-08-12 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Analgesia
Keywords: analgesia; analgesia based sedation; critical care; fentanyl; propofol; remifentanil; sedation; mechanical ventilation; efficacy; safety
MeSH Terms: conditions — Agnosia | interventions — Remifentanil; Injections; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remifentanil (Experimental): Remifentanil analgesia combined with propofol sedation. Treatment was started in patients with an CPOT score of 2 or greater after completion of baseline assessments. All patients received an initial infusion of blinded opioid (placebo bolus dose(6ml) + 6ug/kg per hour infusion at 6 ml/hour). Optimal analgesia (CPOT score ≤2) was then targeted by titrating the infusion in 1.5 ml/hour increments (placebo bolus dose + 1.5ug/kg per hour rate increase).
  Interventions: Drug: Remifentanil
- Fentanyl (Active Comparator): Fentanyl analgesia combined with propofol sedation. Treatment was started in patients with an CPOT score of 2 or greater after completion of baseline assessments. All patients received an initial infusion of blinded opioid (1ug/kg bolus(6ml) + 1ug/kg per hour infusion at 6ml/hour). Optimal analgesia (CPOT score ≤2) was then targeted by titrating the infusion in 1.5 ml/hour increments (1ug/kg bolus dose + 0.25ug/kg per hour rate increase).
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Remifentanil — Dosage forms and strengths: 3 mL Vial/1 mg lyophilized powder. Manufacturer: Yichang Humanwell Pharmaceutical Co.,Ltd
  Other Names: Remifentanil Hydrochloride for Injection
  Arms: Remifentanil
Drug: Fentanyl — Dosage forms and strengths: 50 mcg/mL Fentanyl base/10 mL ampules. Manufacturer: Yichang Humanwell Pharmaceutical Co.,Ltd
  Other Names: Fentanyl Citrate Injection
  Arms: Fentanyl

SUMMARY:
Remifentanil has been approved by the FDA for continuation as an analgesic into the immediate postoperative period in adult patients under the direct supervision of an anesthesia practitioner in a postoperative anesthesia care unit or intensive care setting. However, National Medical Products Administration(NMPA) did not approve this indication. Therefore, the purpose of this study is to confirm the efficacy and safety of remifentanil in the analgesic therapy of critical ill patients in China.

DETAILED DESCRIPTION:
The study was conducted in accordance with good clinical practice and with the guidelines set out in the Declaration of Helsinki. After approval from local and national ethics committees, patients from 17 centres in China were recruited. All patients were randomized, in a double-blind manner, to receive either a remifentanil-propofol regimen or a fentanyl-propofol regimen for analgesia and sedation in the ICU. The aim of the study was to achieve optimal sedation and patient comfort by maintaining an optimal Critical Care Pain Observation Tool (CPOT) score of 2, without clinically significant pain, until the start of the extubation process or for 72 hours, whichever occurred first. CPOT scoring criteria: Facial expressions(Relaxed, neutral=0; Tense=1; Grimacing=2); Body movements(Absence of movements or normal position=0; Protection=1; Restlessness/Agitation=2); Muscle tension(Relaxed=0; Tense, rigid=1; Very tense or rigid=2); Compliance with the ventilator or Vocalization(Tolerating ventilator or movement/Talking in normal tone or no sound=0; Coughing but tolerating/Sighing, moaning=1; Fighting ventilator/Crying out, sobbing=2).

ELIGIBILITY:
Inclusion Criteria:

* Invasive mechanical ventilation with endotracheal intubation
* Expected to continue mechanical ventilation for more than 12 hours
* Informed consent/assent was obtained from all patients or their representatives

Exclusion Criteria:

* Patients with a history of allergy to opioids, benzodiazepines, propofol, or alcohol/drug abuse were excluded from the study
* Patients who are known or suspected to be allergic to the study drug
* Patients whose expected survival time is less than 48h
* Patients receiving deep sedation (RASS≥-4)
* Patients using neuromuscular blocking agent
* Patients who cannot be assessed by RASS
* Patients with myasthenia gravis
* patients with bronchial asthma
* patients with abdominal compartment syndrome
* Patients who need surgery or tracheotomy during the study drug treatment period
* Women during pregnancy and lactation
* Patients who have used short-acting non-steroidal anti-inflammatory drugs within 6 hours
* Patients who have used long-acting non-steroidal anti-inflammatory drugs within 12 hours
* Patients with a history of chronic pain for more than 3 months or who are receiving regular analgesia for more than 3 months
* Patients who have used monoamine oxidase inhibitors within two weeks
* Patients who participate in any clinical trials as subjects within 1 month
* Patients with a history of drug abuse, drug abuse, alcohol abuse* and long-term use of psychotropic drugs within 2 years Alcoholism: Drinking more than 14 times/week (1 time=150ml wine or 360ml beer or 45ml spirits)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2021-06-10 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
analgesia success rate(the proportion of subjects with successful analgesia to the number of subjects in each group) | From study drug administration to actual extubation , up to 72 hours
  Analgesia success is defined as: 1. No salvage analgesics were used during the administration of the study drug; 2 During the administration of the study drug, the time for the analgesia score of subjects to reach the standard (CPOT score ≤ 2) was greater than 70%. CPOT scoring criteria: Facial expressions(Relaxed, neutral=0; Tense=1; Grimacing=2); Body movements(Absence of movements or normal position=0; Protection=1; Restlessness/Agitation=2); Muscle tension(Relaxed=0; Tense, rigid=1; Very tense or rigid=2); Compliance with the ventilator or Vocalization(Tolerating ventilator or movement/Talking in normal tone or no sound=0; Coughing but tolerating/Sighing, moaning=1; Fighting ventilator/Crying out, sobbing=2).

SECONDARY OUTCOMES:
During the study drug administration period, the subjects are in the proportion of optimal time(CPOT score≤2) | From study drug administration to actual extubation , up to 72 hours
  CPOT scoring criteria: Facial expressions(Relaxed, neutral=0; Tense=1; Grimacing=2); Body movements(Absence of movements or normal position=0; Protection=1; Restlessness/Agitation=2); Muscle tension(Relaxed=0; Tense, rigid=1; Very tense or rigid=2); Compliance with the ventilator or Vocalization(Tolerating ventilator or movement/Talking in normal tone or no sound=0; Coughing but tolerating/Sighing, moaning=1; Fighting ventilator/Crying out, sobbing=2).
The number of times the remedial sedative drug propofol was used | From study drug administration to actual extubation , up to 72 hours
  Use the total times of propofol
The proportion of subjects using the salvage sedative drug propofol | From study drug administration to actual extubation , up to 72 hours
  The proportion of subjects who using the salvage sedative drug propofol to the total subjects.
The dosage of the remedial sedative drug propofol | From study drug administration to actual extubation , up to 72 hours
  Use the total dose of propofol
Wearing time from mechanical ventilation | From study drug administration to wearing from mechanical ventilation, up to 72 hours
  Wearing time criteria: The primary disease is improved, and there is no new disease; no use of vasopressors or continuous application of sedative drugs; cough reflex during sputum suction; PEEP≤5cmH2O; PaO2/FiO2≥200mmHg; Minute ventilation<15L/min; 2-minute spontaneous breathing test and passed.
Extubation time | From the start of the extubation process until actual extubation , up to 72 hours
  The start of the extubation process until actual extubation
The success rate of wearing mechanical ventilator | From study drug administration to actual extubation , up to 72 hours
  The proportion of subjects who successfully wearing from mechanical ventilator to the total subjects.
Duration of study drug use in ICU | From study drug administration to the time discharge ICU , up to 72 hours
  The time from the start of the study drug administration to the time discharge ICU.
The proportion of subjects discharging the ICU | From study drug administration to the time discharge ICU, up to 24 weeks
  The proportion of subjects who discharge ICU to the total subjects.
ICU mortality | From study drug administration to the time discharge ICU, up to 24 weeks
  The proportion of subjects who died during ICU admission to the total subjects.
Hospital mortality | From study drug administration to the time discharge hospital, up to 24 weeks
  The proportion of subjects who died during hospital admission to the total subjects.
Length of ICU stay | From administration to discharge ICU, up to 24 weeks
  The number of days the subject stayed in the ICU
Length of hospital stay | From administration to discharge hospital, up to 24 weeks
  The number of days the subject stayed in the hospital
The incidence of study drug-related Lower blood pressure | From study drug administration to actual extubation , up to 72 hours
  Lower blood pressure: mean arterial pressure (MAP) drops more than 25% from the baseline level or requires additional vasopressors;
The incidence of study drug-related slow heart rate | From study drug administration to actual extubation , up to 72 hours
  Slow heart rate: HR<40bpm for less than 1 minute or HR<60 bpm for more than 1 minute;
The incidence of study drug-related respiratory depression | From study drug administration to actual extubation , up to 72 hours
  Respiratory depression: RR<10 bpm or SpO2<90%
Analysis of the cost-effectiveness between remifentanil and fentanyl | From study drug administration to actual extubation , up to 72 hours
  cost-effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: Yang Yi, MD, Study Chair — Department of Critical Care Medicine, Zhongda Hospital, School of Medicine, Southeast University
Locations (17):
- China (17):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Qingyuan People's Hospital, Qingyuan, Guangdong
  - Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Enshi Tujia and Miao Autonomous Prefecture Central Hospital, Enshi, Hubei
  - Yichang Central People's Hospital, Yichang, Hubei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Nanjing Zhong-Da Hospital, Southeast University, Nanjing, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No